CLINICAL TRIAL: NCT00001289
Title: Clinical and Biochemical Effects of Macrophage-Targeted Glucocerebrosidase on Neurological Involvement in Neuronopathic Gaucher's Disease
Brief Title: Effects of Enzyme Replacement in Gaucher's Disease
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 910225; 91-N-0225
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-03-03

CONDITIONS: Gaucher's Disease
Keywords: Enzyme Replacement; Type 3 Gaucher's Disease; Lysosomal Storage; Supranuclear Gaze Palsy; Seizures; Mental Retardation; Gaucher Disease
MeSH Terms: conditions — Gaucher Disease; Seizures; Intellectual Disability

SUMMARY:
Gaucher disease is a lysosomal storage disease resulting from glycocerebroside accumulation in macrophages due to a genetic deficiency of the enzyme glucocerebrosidase. It may occur in adults but occurs most severely in infants, in whom cerebroside also accumulates in neurons. Patients with Gaucher's disease experience enlargement of the liver and spleen and bone destruction. The condition is passed from generation to generation through autosomal recessive inheritance. There are actually three types of Gaucher's disease.

Type I is the most common form. It is a chronic non-neuronopathic form, meaning the disease does not affect nerve cells. The symptoms of type I can appear at any age.

Type II appears in infancy and usually results in death for the patient. Type II is an acute neuronopathic form and can affect the brain stem. It is the most severe form of the disease.

Type III is also neuronopathic, however it is subacute in nature. This means the course of the illness lies somewhere between long-term (chronic) and short-term (acute).

The purpose of this study is to examine the effects of enzyme replacement therapy on patients with Gaucher's disease, specifically those types directly affecting the nervous system (neuronopathic).

Patients with Gaucher's disease types II and III will be selected to participate in the study and receive enzyme replacement therapy. Patients participating will undergo a variety of tests to measure levels of hemoglobin concentration, liver volume, and spleen volume. Improvements in these measures will be compared other laboratory tests measuring the involvement of the nervous system.

DETAILED DESCRIPTION:
The purpose of this study is to examine the effects of enzyme replacement therapy in patients with neuronopathic Gaucher's disease and to investigate the pathogenesis of their neurological signs and symptoms. Macrophage-targeted glucocerebrosidase will be administered by intravenous infusion under the supervision of the patient's private physician at an initial dosage of 60 to 120 IU per kg of body weight weekly or every other week. Patients will be categorized as treatment responders if they display a clinically significant increase in hemoglobin concentration and a reduction in hepatic or splenic volume. Improvement in these parameters over time will be correlated with measurements for metabolic encephalopathy and radiologic, electrophysiologic and psychometric measurements of neurological involvement.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. All patients with neuropathic Gaucher's disease who have a partial or complete horizontal supranuclear gaze palsy or a genotype associated with neurological involvement.
  2. All candidates must be serologically nonreactive for hepatitis B and human immunodeficiency (AIDS) virus. HIV positive patients will be excluded because of the effects of the latter illness on cognitive performance.
  3. Individuals with neoplastic disease will be excluded.
  4. The general health and well being of each candidate must be sufficient to allow for a modest amount of blood drawing, collection of appropriate urine and spinal fluid specimens and performance of necessary roentgenographic and magnetic resonance (MR) imaging studies. In addition, each candidate must be able to return to the National Institutes of Health (NIH) on a regular basis dictated by disease severity for monitoring of laboratory parameters.

EXCLUSION CRITERIA:

1. Patient who participates in a clinical study of an investigational therapeutic agent for Gaucher Disease.
2. Patient and/or the patient's parent(s) or legal guardian(s) are unable to understand the nature, scope, and possible consequences of the study.
3. Patient is unable to comply with the protocol, e.g., uncooperative with protocol schedule, refusal to agree to all of the study procedures.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70
Dates: Start 1991-09-23; Study Completion 2008-03-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Barton NW, Brady RO, Dambrosia JM, Di Bisceglie AM, Doppelt SH, Hill SC, Mankin HJ, Murray GJ, Parker RI, Argoff CE, et al. Replacement therapy for inherited enzyme deficiency--macrophage-targeted glucocerebrosidase for Gaucher's disease. N Engl J Med. 1991 May 23;324(21):1464-70. doi: 10.1056/NEJM199105233242104. PMID 2023606
- [Derived] Benko W, Ries M, Wiggs EA, Brady RO, Schiffmann R, Fitzgibbon EJ. The saccadic and neurological deficits in type 3 Gaucher disease. PLoS One. 2011;6(7):e22410. doi: 10.1371/journal.pone.0022410. Epub 2011 Jul 20. PMID 21799847